CLINICAL TRIAL: NCT04619706
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase IIA Study of FSD201 (Ultramicronized PEA) + Standard of Care (SOC) Vs SOC in the Treatment of Hospitalized Patients With COVID-19
Brief Title: Ultramicronized Palmitoylethanolamide (PEA) Treatment in Hospitalized Participants With COVID-19
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties recruiting new subjects
Sponsor: Quantum Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FSD201-03
Record Dates: First submitted 2020-11-05; First posted 2020-11-06 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: FSD201 600 mg (Experimental): Participants will receive 600 milligrams (mg) FSD201 tablet twice daily (BID) orally along with the placebo matched to 600 mg FSD201 tablet from Day 1 to Day 14.
  Interventions: Drug: FSD201; Drug: Placebo; Other: Standard of Care for Covid-19
- Arm B: FSD201 1200 mg (Experimental): Participants will receive 1200 mg (2x600 mg) tablets FSD201 BID orally from Day 1 to Day 14.
  Interventions: Drug: FSD201; Other: Standard of Care for Covid-19
- Arm C: Placebo (Placebo Comparator): Participants will receive placebo matched to 600 mg FSD201 tablets (2xplacebo tablets) from Day 1 to Day 14.
  Interventions: Drug: Placebo; Other: Standard of Care for Covid-19

INTERVENTIONS:
Drug: FSD201 — Tablets for oral administration.
  Other Names: ultramicronized palmitoylethanolamide (PEA)
  Arms: Arm A: FSD201 600 mg; Arm B: FSD201 1200 mg
Drug: Placebo — Placebo tablets matched to FSD201 for oral administration.
  Arms: Arm A: FSD201 600 mg; Arm C: Placebo
Other: Standard of Care for Covid-19 — Standard of care for Covid-19 as determined by site PI

SUMMARY:
This study will measure the effect of FSD201 (ultramicronized PEA) + SoC vs placebo + SoC on Day 28, on disease progression in the confirmed coronavirus disease 2019 (COVID-19) patient population.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing and able to give informed consent to participate in the study
* Has admitted to a hospital and has a positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test by standard reverse transcription-polymerase chain reaction (RT-PCR) assay or equivalent test
* Has the presence of any symptom(s) suggestive of moderate or severe systemic illness with COVID-19 on Day 1 such as the presence of fever (greater than or equal to (>=)38.0 degree Celsius [>=100.4 degree fahrenheit] by any route), "feeling hot," "feeling sweaty," headache, malaise, fatigue, muscle pain, diarrhea, nausea, vomiting, cough, sore throat, or shortness of breath upon exertion and/or at rest, or respiratory distress
* Has the presence of moderate to severe clinical signs indicative of moderate or severe illness with COVID-19 on Day 1. A. Moderate: (1) Clinical signs suggestive of moderate illness with COVID-19, such as respiratory rate >=20 breaths per minute, SpO2 >93% on room air at sea level, heart rate >=90 beats per minute. (2) No clinical signs indicative of severe or critical COVID-19. B. Severe: (1) Clinical signs suggestive of severe systemic illness with COVID-19, such as respiratory rate >=30 breaths per minute, heart rate >=125 beats per minute, SpO2 less than or equal to (<=) 93% on room air at sea level or partial pressure of oxygen (PaO2)/fraction of inspired oxygen (FiO2) less than (<)300, heart rate >=125 beats per minute. (2) No criteria met for critical COVID-19
* Has either normal renal function or mild or moderate renal impairment: estimated creatinine clearance >30 milliliters per minute (mL/min) on Day 1
* Able to swallow the study drug (tablets)
* Men whose sexual partners are women of childbearing potential (WOCBP) must agree to comply with one of the following contraception requirements from the time of first dose of study medication (Day 1) until at least 30 days after the last dose of study medication: (a) Vasectomy with documentation of azoospermia. (b) Sexual abstinence. (c) Male condom plus partner use of one of the contraceptive
* WOCBP must agree to comply with one of the following contraception requirements from the time of first dose of study medication (Day 1) until at least 30 days after the last dose of study medication: (a) Sexual abstinence (b) Use of one of the contraceptive options (c) Vasectomy of male partner with documentation of azoospermia

Exclusion Criteria:

* The participant, in the opinion of the investigator, is not likely to survive for >=48 hours beyond Day 1
* Has a diagnosis of asymptomatic COVID-19, mild COVID-19, or critical COVID-19 on Day 1
* Has a documented current liver disease, or known hepatic or biliary abnormalities (with the exception of asymptomatic gallstones) at screening or on Day 1
* Has a Child Pugh score >= C
* Has a documented medical history of infection with human immunodeficiency virus or hepatitis A, B, or C at screening or on Day 1
* Has a documented active infection with tuberculosis at screening or on Day 1
* Has clinically significant ECG abnormalities at screening or on Day 1
* Requires dialysis or is on any renal replacement therapies at screening or on Day 1
* A female participant who is pregnant or planning to become pregnant during the study, breastfeeding, or has a positive pregnancy test at screening
* Receiving alpha-blockers, combined alpha/beta blockers, antihistamines, or any drugs that will affect the levels of cytokines released due to immune stress
* Has received any immunoglobulins within 6 months of screening or planned administration of any immunoglobulins during the screening and/or treatment periods
* Has a known history of drug abuse within 6 months of study start that would interfere with the participant's participation in the study
* Has a history of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, would contraindicate their participation
* Has participated in and/or plan to participate in another clinical study
* Will be transferred to another hospital which is not a study site within 72 hours
* Cannot read and speak either English or Spanish

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Disease Progression at Day 28 | Day 28
  Disease progression will be defined as the percentage of participants who are not alive or who have respiratory failure. Respiratory failure will be defined as the need for invasive or non-invasive mechanical ventilation, high-flow oxygen, or extracorporeal membraneoxygenation (ECMO).

SECONDARY OUTCOMES:
Percentage of Participants With Disease Resolution at Day 28 | Day 28
  Disease resolution will be defined as participants alive and not requiring supplemental oxygen (at home or in the hospital).
Percentage of Participants Requiring Invasive Mechanical Ventilation or ExtraCorporeal Membrane Oxygenation (ECMO) or who are not Alive on Day 28 | Day 28
Change From Baseline in Oxygen use | Baseline, Day 15, and Day 28
  Oxygen use will be assessed by change in the type of oxygen use between the following categories: no oxygen, supplemental oxygen, non-invasive mechanical ventilation or high-flow oxygen, invasive mechanical ventilation/ECMO.
Change From Baseline in Saturation of Oxygen (SpO2) percent (%) | Baseline through Day 28
Change From Baseline in Clinical Status Related to COVID-19 | Baseline, Day 15, and Day 28
  Clinical status will be measured with the 9-point ordinal scale ranging (1-9; 1 being death and 9 being not hospitalized, not requiring supplemental home oxygen, and no limitations on activities).
Percentage of Participants who Die (Mortality Rate) at Day 28 | Day 28
  Mortality rate will be defined as the percentage of participants who die.
Percentage of Participants Testing Negative for COVID-19 at Day 28 | Day 28
  COVID-19 testing by standard standard reverse transcription-polymerase chain reaction (RT-PCR) assay or equivalent test.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the signing of the informed consent to Day 60 (approximately 9 months)
  Number of participants with AEs and SAEs will be summarized and reported by seriousness, severity, relationship to the study medication, outcome, and duration.
Number of Participants With Clinically Significant Changes in Vital Signs, Laboratory Parameters, Electrocardiogram Findings and Physical Examination Findings | Baseline through Day 28
  The number of participants with clinically significant changes in vital signs, laboratory parameters and electrocardiogram findings, and physical findings will be reported.
Plasma Concentrations of FSD201 | Day 1 and Day 14
  Plasma concentrations will be measured in participants who give optional consent will be collected relative to the first dose on Day 1 and the first dose on Day 14. Samples on Day 1 and Day 14 will be collected predose (within 10 minutes before the first daily dose) and post dose at 2 hours (±30 minutes), 12 hours (±30 minutes) (before the evening dose), and 24 hours (±30 minutes)(before the next morning dose).
Maximum Observed Plasma Concentration (Cmax) of FSD201 | Day 1 and Day 14
  Cmax is defined as maximum observed plasma concentration.
Area Under the Concentration-Time Curve (AUC) of FSD201 | Day 1 and Day 14
  Area under the concentration-time curve (AUC).
Elimination Half-Life (t1/2) | Day 1 and Day 14
  Elimination half-life (t1/2) of FSD201.
Apparent Total Body Clearance (CL/F) of FSD201 | Day 1 and Day 14
  CL/F is the apparent total body clearance of FSD201 in plasma.
Apparent Volume of Distribution (Vz/F) of FSD201 | Day 1 and Day 14
  Vz/F is the apparent volume of distribution of FSD201 in plasma.
Average Observed Plasma Concentration at Steady State (Cav) of FSD201 | Day 1 and Day 14
  Cav is average plasma concentration over a dosing interval.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Miami, Florida, Miami, Florida
  - Palms of Pasadena Hospital, Saint Petersburg, Florida, St. Petersburg, Florida
  - Theia Clinical Research, St. Petersburg, Florida, St. Petersburg, Florida
  - Idaho Falls, Idaho, Idaho Falls, Idaho
  - Winfield, Illinois, Winfield, Illinois
  - Butte, Montana, Butte, Montana
  - Tulsa, Oklahoma, Tulsa, Oklahoma
  - Kingsport, Tennessee, Kingsport, Tennessee
  - Amarillo, Texas, Amarillo, Texas
  - Mesquite, Texas, Mesquite, Texas

IPD SHARING:
Plan to Share IPD: No